CLINICAL TRIAL: NCT06527976
Title: Dexmedetomedine Versus Dexamethasone in Ultrasound Guided Adductor Canal Block for Patients Undergoing Knee Arthroscope
Brief Title: Dexamethasone Versus Demedetomidine Addition for Adductor Canal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, Asisstant professor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12222
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomedine added to bupivacaine for adductor canal block
  Arms: dexmedetomidine
Drug: Dexamethasone — dexamethasone added to bupivacaine for adductor canal block
  Arms: dexamethasone

SUMMARY:
Single-injection peripheral nerve block (PNB) is commonly used for perioperative analgesia and anesthesia. Three approaches for extending the duration of PNB include continuous PNB with catheter-based techniques, novel local anesthetics delivery systems and addition of novel adjuvants to local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* elective operation
* ASA STATUS I and II

Exclusion Criteria:

* patient refusal
* ASA status III and IV
* contraindications to local anesthesia

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
visual analogue scale score | 24 hours postoperative
  scale of 11 points. zero=no pain, 10 = worest pain ever

SECONDARY OUTCOMES:
analgesia duration | 24 hours postoperative
  pain free duration after block
opioid consumption | 24 hours postoperative
  amount of opioid consumed postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt